CLINICAL TRIAL: NCT02196597
Title: Prospective Multi-center Evaluation of the Value of Anorectal Manometry Before Closure of Protective Ileostomy or Sigmoidostomy After Rectal Resection in Patients With Rectal Carcinoma
Brief Title: Value of Anorectal Manometry Before Ileo- or Sigmoidostomy Closure After Rectal Resection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: German Society for Neurogastroenterology and Motility (Other)
Responsible Party: Principal Investigator, Dr. Christian Pehl, Chairman, German Society for Neurogastroenterology and Motility
Other Study IDs: DGNM_ARM
Record Dates: First submitted 2013-11-04; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Fecal Incontinence; Quality of Life
Keywords: anorectal manometry
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- resection with RCT: rectal resection in the case of rectal carcinoma with preoperative radiochemotherapy
- resection without RCT: patients with rectal resection without preoperative radiochemotherapy

SUMMARY:
Background: High prevalence of fecal incontinence after rectal resection in patients with rectal carcinoma.

Hypothesis: Anorectal manometry done before ileostomy or sigmoidostomy closure can predict fecal incontinence.

Methods: Anorectal manometry before, 1 month and 6 month after closure. Anorectal endosonography before and 1 month after closure. Prediction of postoperative incontinence by the surgeon (digital sphincter examination). Visual analog scales for continence, subjective success of operation, and global well being; Wexner and Vaizey incontinence score; Parks incontinence classification; Rockwood fecal incontinence quality of life score; each before, 1 and 6 month after closure.

ELIGIBILITY:
Inclusion Criteria:

* all patients planned for ileo- or sigmoidostomy closure after rectal resection for rectal carcinoma

Exclusion Criteria:

* preoperative incontinence for solid stool
* dementia
* pregnancy
* latex allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients operated for rectal carcinoma in three German centers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
predictive value of preoperative anorectal manometry for postoperative fecal incontinence | 6 month postoperative
  Anorectal manometry is done preoperatively. Fecal incontinence is determined at 6 month postoperatively. Analysis of correlation between preoperative manometry parameter and incidence of postoperative fecal incontinence.

SECONDARY OUTCOMES:
fecal incontinence in patients with/without neoadjuvant radiochemotherapy | six month postoperative
  Comparison of the percentage of patients with postoperative fecal incontinence after rectal resection in patients with or without neoadjuvant radiochemotherapy
predictive value of the surgeon's preoperative evaluation | six month postoperative
  Clinical evaluation of the patient preoperatively with estimation (written statement) about postoperative continence/incontinence. Fecal incontinence is determined at 6 month postoperatively. Analysis of correlation between the surgeons´ predictions and the incidence of postoperative fecal incontinence

OTHER OUTCOMES:
prediction of postoperative fecal incontinence by the score of Stadelmaier and Matzel (Score =18.230 - 0.94x anastomotic level - 0.18 x resting pressure + 3.72 x radiochemotherapy (done 1, not done 0) | six month postoperative
  Analysis of correlation between the preoperatively predicted Wexner score and the observed Wexner score six month postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Pehl, MD, Principal Investigator — German Society for Neurogastroenterology and Motility
Locations (3):
- Germany (3):
  - Hosptial Landshut-Achdorf, Landshut
  - Hospital Memmingen, Memmingen
  - Hospital Vilsbiburg, Vilsbiburg

REFERENCES:
- [Result] Stadelmaier U, Bittorf B, Meyer M, Hohenberger W, Matzel KE. [Can continence function after rectal resection be prognostically estimated?]. Chirurg. 2000 Aug;71(8):932-8. doi: 10.1007/s001040051158. German. PMID 11013813
- See also: Homepage of the German Society for Neurogastroenterology and Motility — http://www.neurogastro.de